CLINICAL TRIAL: NCT03952286
Title: ED-Initiated School-based Asthma Medication Supervision
Acronym: EDSAMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1R34HL137851 (NIH)
Record Dates: First submitted 2019-05-03; First posted 2019-05-16 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2022-05

CONDITIONS: Asthma; Asthma in Children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Group 1 receives the intervention: ED-Initiated School-based Asthma Medication Supervision (school and home asthma medication supervision). Group 2 receives usual care (home asthma medication supervision).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): ED-Dispensing with home and school supervision
  Interventions: Drug: ED-Dispensing home and school supervision
- Control (Other): ED-Dispensing with home supervision
  Interventions: Drug: ED-Dispensing home and school supervision

INTERVENTIONS:
Drug: ED-Dispensing home and school supervision — 1. Oral prednisolone based on body weight to achieve a daily dose of 2mg/kg/day not to exceed 40 mg per day for 5 days or its equivalent (provided in the emergency department),
  2. 360 ug of budesonide inhalation powder once-daily for at-home use, and
  3. albuterol sulfate as needed for relief of acute respiratory symptoms.

SUMMARY:
Asthma is a common chronic condition that causes substantial morbidity among children and much of it is attributable to medication non-adherence. The National Asthma Education and Prevention Program (NAEPP) and the American Academy of Asthma, Allergy, and Immunology have urged others to develop more effective adherence programs.Schools are a logical setting to deploy such interventions because they are where children congregate, spend much of their day, and are frequently monitored. Because many schools serve a high proportion of minority and low-income students, engaging them presents a unique opportunity to reach populations who experience the greatest burden of preventable morbidity.

Supervising inhaled corticosteroid (ICS) use in the school setting can increase medication adherence and reduce episodes of poor asthma control. Under certain conditions, it can also be cost-effective. However, recruiting children from school settings tends to enroll children with mild asthma and infrequent health care use. Therefore, initiating supervised treatment in these children tends to burden school personnel with unnecessary work and diminishes the program's cost-effectiveness. To address this inefficiency, the investigators propose to recruit children who are discharged from the Hospital Emergency Departments (EDs) following successful treatment of an asthma attack. Such children have much higher risk of a future asthma attack than their peers.

The Pediatric Emergency Care Applied Research Network (PECARN) com- prises10 hospital-affiliated EDs that serve 1 million acutely ill and injured children annually. Their primary research mission is to reduce childhood morbidity and mortality by establishing creative partnerships between emergency medical service providers and their surrounding communities. The networks size and geographic diversity make it uniquely situated to develop, implement, and evaluate the feasibility and effectiveness of ED-Initiated School-Based Asthma Medication Supervision (ED-SAMS).

Approximately one-third of children treated for an asthma attack within PECARN experience a second ED-managed attack within 6 months. While the NAEPP guidelines recommend that long-term ICS treatment should be initiated at ED discharge, <20% of children actually receive a prescription for controller therapy. Observational data indicate that patients who use ICS following discharge are almost half as likely as non-users to experience a repeat ED visit. Many have also argued that ED-initiated treatment could be cost-effective. However, simply providing patients with a prescription does not ensure that they will actually use it once discharged. To ensure better medication adherence, the investigators propose to dispense ICS at discharge and supervise its use in the school setting.

DETAILED DESCRIPTION:
Approximately 8% of children in the United States have asthma. Each year, these children experience 4 million asthma attacks that result in 725,000 ED visits and 100,000 hospitalizations. Unsurprisingly, the direct medical expenditures of children with asthma are 75-90% higher than those of children without asthma. In 2016, this amount totaled 40 billion dollars. Substantial indirect costs are incurred when parents miss work to care for their children who miss school. These additional costs raise the total economic burden of asthma to $80 billion annually. Frequent asthma-related school absences impair academic achievement and social functioning. This burden falls disproportionately on minority, low-income, and urban populations. For example, black children have 60% more ED visits and 75% more hospitalizations than white children even though they have similar asthma attack rates.

Adherence to ICS is notoriously poor.20, 22, 23 While 86% of privately insured patients who receive an ICS prescription will refill it within 30 days, only 64% will subsequently refill it again within 180 days. Even worse, only 3% will refill enough medication to cover greater than or equal to 75% of prescribed days with average medication possession being approximately 20%. Black and Hispanic patients are 20% less likely to refill their initial prescription and are 40% less likely to refill enough medication to cover greater than or equal to 75% of prescribed days. Adherence is similarly poor among the publicly insured. Among Medicaid-insured children, ICS is only refilled enough to cover 20% of prescribed days; fewer than 15% will refill enough to cover greater than or equal to 50% of days. At any given time, 40% of children with asthma are not well-controlled and much of this is attributable to nonadherence. Simulation and modeling studies suggest that maximizing ICS adherence among those prescribed ICS could reduce health care utilization by 25-45%. Even greater reductions are hypothesized if ICS prescribing could be expanded to all patients at risk of serious asthma-related exacerbations. However, a recent Cochrane review concluded that current methods of improving adherence for chronic health problems are mostly complex and not very effective. New adherence strategies will be needed if society is to achieve the gains suggested possible by simulations. Medication non-adherence among patients with chronic disease is a multi-dimensional challenge. The cost and convenience of obtaining medication (health system factors) and the motivation needed to adhere with a daily health habit (patient-related factors) are common barriers to adherence that are addressed by this study. Medication acquisition costs deter patients from refilling and refilling prescription medications. Even small $1-3 co-payments can appreciably reduce adherence. However, imposing additional time costs by requiring more frequent refills has an even greater impact. Time costs can add $50-100 per prescription. Therefore, the $155 out-of-pocket spending estimate for children's asthma medication likely understates the true economic burden. Dispensing ICS in the ED is therefore expected to improve adherence by reducing the substantial time and travel costs associated with medication acquisition. ICS treatment also burdens patients by requiring them to adopt a daily health habit. For children, this burden primarily falls on parents. Parents weigh the perceived benefits of treatment against their perceptions of treatment risk and burden. Given that asthma symptoms fluctuate in response to treatment and season, many purposefully reduce medication administration when their child's symptoms wane (volitional non-adherence).

In the absence of treatment, the underlying inflammation is allowed to worsen and exacerbation risk increases. This reactive pattern of medication use is substantiated by the fact that 37% of all prescriptions for ICS are refilled on the same day as prescriptions for oral corticosteroid, suggesting after the exacerbation, not before it.18 Even more disturbing, less than 50% of children who refilled a prescription for oral corticosteroid were ever noted to have refilled an ICS prescription, meaning most lacked any access to controller medication.18 Our proposal addresses the problem of primary non-adherence by dispensing medication in the ED and addresses non-adherence by arranging supervised use in the school setting.

ELIGIBILITY:
Inclusion Criteria:

1. Children 6-12 years of age; AND
2. Treated for an asthma exacerbation as determined clinically by the principal ED provider based on symptoms such as shortness-of-breath, cough, and wheezing; AND
3. Symptoms must improve following more than 1 dose of albuterol and more than 1 dose of systemic corticosteroids such that he/she can be safely discharged home; AND
4. Must have physician-diagnosed

Exclusion Criteria:

1. Attends a non-participating school; OR
2. Attends a participating school less than 5x/week; OR
3. Enrolled in another research study; OR
4. Patients who are hospitalized; OR
5. The patient or their consenting parent/guardian does not speak English or Spanish; OR
6. ICU admissions for asthma in the past year; OR
7. History of more than 2 hospitalizations for asthma in past year; OR
8. History of more than 2 controller medications for asthma in the past 30 days; OR
9. Study medication represents a step-down in asthma therapy in the judgement of the ED physician; OR
10. Parent does not have a cell phone; OR
11. Parent cannot send and receive text messages.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Asthma & Airway Disease Research Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gerald LB, Gerald JK, VanBuren JM, Lowe A, Guthrie CC, Klein EJ, Morrison A, Startup E, Denninghoff K. Randomized trial of the feasibility of ED-initiated school-based asthma medication supervision (ED-SAMS). Pilot Feasibility Stud. 2021 Sep 27;7(1):179. doi: 10.1186/s40814-021-00913-0. PMID 34579785

RESULTS

PARTICIPANT FLOW:
Groups:
- ED-Dispensing With Home and School Supervision: ED-Dispensing home and school supervision: 1. Oral prednisolone based on body weight to achieve a daily dose of 2mg/kg/day not to exceed 40 mg per day for 5 days or its equivalent (provided in the emergency department), 2. 360 ug of budesonide inhalation powder once-daily for at-home use, and 3. albuterol sulfate as needed for relief of acute respiratory symptoms.
- ED-Dispensing With Home Supervision: ED-Dispensing home supervision: 1. Oral prednisolone based on body weight to achieve a daily dose of 2mg/kg/day not to exceed 40 mg per day for 5 days or its equivalent (provided in the emergency department), 2. 360 ug of budesonide inhalation powder once-daily for at-home use, and 3. albuterol sulfate as needed for relief of acute respiratory symptoms.
Period: Overall Study
Arm/Group | ED-Dispensing With Home and School Supervision | ED-Dispensing With Home Supervision
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ED-Dispensing With Home and School Supervision | ED-Dispensing With Home Supervision | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.2 (0.89) | 8.4 (1.86) | 7.9 (1.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 1 | 1 | 2
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: 90-day Emergency Department (ED) Recidivism
Description: 90-day Emergency Department (ED) Recidivism as measured by the number of participants that return to the ED for asthma exacerbation within 90 days of discharge
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | ED-Dispensing With Home and School Supervision | ED-Dispensing With Home Supervision
Number analyzed (Participants) | 6 | 7
Participants | 1 | 2

2. Secondary Outcome: Cost-effectiveness
Description: Cost-effectiveness as estimated by the dollars per averted ED visit
Time Frame: 90 days
Population: Cost-effectiveness analysis cannot be completed because an estimate of ED days averted was not collected due to low enrollment. Therefore, the cost-effectiveness outcome, which is dollars per averted ED visit, could not be calculated.
Arm/Group | ED-Dispensing With Home and School Supervision | ED-Dispensing With Home Supervision
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | ED-Dispensing With Home and School Supervision | ED-Dispensing With Home Supervision
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT03952286/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03952286/SAP_001.pdf
  • Informed Consent Form (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT03952286/ICF_002.pdf